CLINICAL TRIAL: NCT01971411
Title: Vitamin D Deficiency in Elderly African American Women in Central Texas
Status: Completed | Type: Observational
Sponsor: McLennan County Medical Education and Research Foundation (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: VIT.D.DEF.1
Record Dates: First submitted 2013-04-23; First posted 2013-10-29 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Vitamin D Deficiency; Osteoporosis; Osteopenia
Keywords: Hyperparathyroidism; Hypoparathyroidism; Calcium; Vitamin D; Bone mineral density; African American; Female; Elderly
MeSH Terms: conditions — Vitamin D Deficiency; Osteoporosis; Bone Diseases, Metabolic; Hyperparathyroidism; Hypoparathyroidism | interventions — Calcium; Ergocalciferols; Vitamin D; Magnesium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Community dwelling elderly black females
  Interventions: Drug: Calcium 500mg with 200 IU Vitamin D - 2 tablets daily; Procedure: Blood levels of Vitamin D, Serum CTX, Mg, Ca++ and iPTH; Behavioral: Usual sun exposure documentation; Behavioral: Dietary intake of calcium, vitamin D, magnesium

INTERVENTIONS:
Drug: Calcium 500mg with 200 IU Vitamin D - 2 tablets daily
Procedure: Blood levels of Vitamin D, Serum CTX, Mg, Ca++ and iPTH
Behavioral: Usual sun exposure documentation
Behavioral: Dietary intake of calcium, vitamin D, magnesium

SUMMARY:
In order to make bone health a reality for older adults, we need to consider the prevalence of Vitamin D deficiency in relation to environment latitude as well as vitamin D supplementation. Darker skin pigmentation and aging are known factors influencing the body's ability to synthesis adequate amounts of Vitamin D. The aim of this project is to document vitamin D deficiency in elderly African American women living in a southern latitude.

DETAILED DESCRIPTION:
Summary: Since darker skin pigmentation and aging are known factors influencing the body's ability to synthesis adequate amounts of Vitamin D, we hypothesize that: 1) the usual sun exposure in the southern United States may not be sufficient to maintain adequate vitamin D levels in elderly African American women, 2) recommended supplementation of Vitamin D 400 IU/d may not be adequate to prevent Vitamin D deficiency which in turn could lead to calcium deficiency and possibly sub-clinical hyperparathyroidism.

This study will enroll 60 African American women age 65 or older who do not have renal, hepatic or gastrointestinal disorders that could affect Vitamin D and calcium absorption and metabolism. Patients will have two scheduled office visits. Demographic data will be collected with attention to dietary intake of calcium and vitamin D, and the patient's customary degree of sun exposure. Ca, 25-hydroxyvitamin D, PTH and serum CTX (a bone resorption marker) are measured on enrollment day and repeated 6 weeks later. All patients not already taking 1000 mg Calcium with 400 IU of Vitamin D orally daily were given samples of this supplement to last for 6 weeks without making any change in diet or sun exposure recommendations. The study period will extend April to June - a time when there should be ample sunlight but it is not so hot as to stop the elderly from going outdoors. Statistical analysis will be performed as to the effect(s) of ethnic background, age, diet, and intensity of sun exposure as related to Ca, 25-hydroxyvitamin D, PTH and serum CTX.

ELIGIBILITY:
Inclusion Criteria:

1. Age 70 or older woman
2. African American ethnicity
3. Non-institutionalized

Exclusion Criteria:

1. De-compensated hepatic insufficiency
2. Renal insufficiency with GFR estimated to be < 30 ml/min
3. Gastrointestinal disorders that might affect absorption such as known malabsorption, celiac sprue, short gut or blind loop syndrome.
4. Institutionalized

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: African American females aged 70 years or older and non-institutionalized
Sampling Method: Non-Probability Sample
Enrollment: 60
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 6 week period in 2007

CONTACTS AND LOCATIONS:
Overall Officials: Sally P Weaver, PhD, MD, Principal Investigator — McLennan County Medical Educ. and Research Foundation; H. S. Eugene Fung, MD, Principal Investigator
Locations (1):
- Family Practice Center, Waco, Texas, United States

REFERENCES:
- [Result] Weaver SP, Passmore C, Collins B, Fung E. Vitamin D, sunlight exposure, and bone density in elderly African American females of low socioeconomic status. Fam Med. 2010 Jan;42(1):47-51. PMID 20063223